CLINICAL TRIAL: NCT05488366
Title: A Pilot Study of Immunotherapy Combined With Stereotactic Ablative Radiotherapy for Patients With Advanced or Metastatic Sarcoma
Brief Title: Immunotherapy Combined With Radiotherapy for Metastatic Sarcoma
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Jeremy Harris, Assistant Clinical Professor, University of California, Irvine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCI 21-03 [HS# 978]; 978 (Other: University of California, Irvine)
Record Dates: First submitted 2022-08-01; First posted 2022-08-04 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Sarcoma, Soft Tissue
Keywords: Sarcoma; Advanced Sarcoma; Metastatic Sarcoma; Pembrolizumab; Stereotactic Ablative Radiotherapy
MeSH Terms: conditions — Sarcoma | interventions — pembrolizumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- A: Pembrolizumab + Radiation Therapy (Experimental): Patients receive pembrolizumab 400 mg intravenous every 42 days; Radiation therapy in 1 to 10 fractions.
  Interventions: Drug: Pembrolizumab; Radiation: Radiation therapy
- B: Radiation Therapy with or without standard of care checkpoint inhibitor immunotherapy (Experimental): Patients who are currently receiving a checkpoint inhibitor immunotherapy regimen will be allowed to continue their regimen at their treating oncologist's discretion. Radiation therapy will be delivered in 1 to 10 fractions starting on Day 1.
  Interventions: Radiation: Radiation therapy

INTERVENTIONS:
Drug: Pembrolizumab — Given IV
  Other Names: MK-3475
  Arms: A: Pembrolizumab + Radiation Therapy
Radiation: Radiation therapy — Single target will be selected by the treating radiation oncologist. A lesion causing symptoms or expected to become symptomatic will be favored for target selection.
  Other Names: RT

SUMMARY:
This is a pilot study determining the feasibility of combination treatments, pembrolizumab and stereotactic ablative radiotherapy (SBRT) in subjects with soft-tissue sarcoma. These are subjects who have metastatic disease initially, or recurrent or progressive disease that is not eligible for curative surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed soft-tissue sarcoma, or a soft-tissue sarcoma with tumor mutational burden ≥10 mut/Mb.
* Patient must either have started a checkpoint inhibitor immunotherapy regimen within 60 days, or have a soft-tissue sarcoma histology amenable to pembrolizumab therapy (inclusive of undifferentiated pleomorphic sarcoma [formerly known as malignant fibrous histiocytoma], myxofibrosarcoma, dedifferentiated liposarcoma or undifferentiated sarcoma [unclassified histology]).
* Patients with soft-tissue sarcoma must have advanced disease (stage IV) or previously treated disease that has become progressive, recurrent, or metastatic, and either previously received first-line systemic therapy or been deemed ineligible to receive first-line systemic therapy. Staging is by AJCC 8th Edition.
* Must not have disease amenable to curative intent surgery.
* Must have at least 2 measurable lesions per RECIST v1.1 assessed by CT scan. A measurable lesion is defined to mean at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >20 mm with conventional techniques or as >10 mm with spiral CT scan.
* Must have at least 1 site of non-central nervous system (CNS) disease amenable to treatment with radiation therapy. This lesion may have been previously treated with radiation if the cumulative spinal cord dose will remain below a Biologically Effective Dose (BED)α/β 2Gy of 112 Gy (single fraction equivalent 14 Gy) and the radiation will be delivered at least 180 days after completion of the prior radiation course to the same site. BED will be calculated using the linear-quadratic formula: d * f * (1 + [d / (α/β)]), where d is the dose per fraction, f is the total number of fractions, and α/β is the property of irradiated tissue measured in Gray.
* Must be age ≥ 18 years. Because initial and subsequent therapies for pediatric sarcomas (<18 years of age) are different than those ≥18, children are excluded from this study. In addition, because no adverse event data are currently available on the use of SBRT combined with pembrolizumab in patients <18 years of age, children are excluded from this study but will be eligible for future pediatric trials, if applicable.

  1. Both men and women and members of all races and ethnic groups are eligible for this trial. Non-English speaking, deaf, hard of hearing and illiterate individuals are eligible for this trial
* Performance status: ECOG performance status ≤2 (Karnofsky ≥50%).
* Life expectancy of ≥3 months.
* Adequate organ and marrow function as defined below. Labs should be performed within 14 days of treatment.

  1. Leukocytes ≥2,000/mcL
  2. Absolute neutrophil count ≥1,000/mcL
  3. Platelets ≥75,000/mcL
  4. AST(SGOT)/ALT(SPGT) ≤3 times institutional upper limit of normal (ULN), or ≤5 times ULN for patients with liver metastases
  5. Total bilirubin ≤2.5 times institutional ULN
  6. Serum creatinine ≤2.5 times institutional ULN, or calculated creatinine clearance ≥30 mL/min (if serum creatinine >2.5 times institutional ULN)
  7. Thyroid stimulating hormone within institutional limits, or T4 is within institutional limits if TSH is outside of institutional limits
* Female patients of childbearing potential must have a negative urine or serum pregnancy within 72 hours before receiving the first dose of pembrolizumab. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* The effects of pembrolizumab and ionizing radiation on the developing human fetus are known to have the potential for congenital abnormalities and fetal harm. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 120 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

  1. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
  1. Has not undergone a hysterectomy or bilateral oophorectomy; or
  2. Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Patients who are HIV-positive with undetectable HIV viral load are eligible provided they meet all other protocol criteria for participation.
* Patients with HBV or HCV infection are eligible provided viral loads are undetectable. Patients on suppressive therapy are eligible.
* Patients must not be on active immunosuppression within 7 days prior to the first dose of treatment.
* Patients must not have a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 2 weeks prior to initiation of study therapy.
* Patients who have not recovered from adverse events due to prior anti-cancer therapy administered.
* Patients must not be receiving any other investigational agents.
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to pembrolizumab.
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.

  1. Pembrolizumab can cause fetal harm when administered to a pregnant woman based on the biological mechanism that PD-1/PD-L1 signaling is an important pathway in the maintenance of pregnancy through induction of maternal immune tolerance to fetal tissue.1 Human IgG4 is known to cross the placenta. Animal models have found that blocking PD-L1 signaling increases the risk of fetal loss, and immune-mediated disorders occurred in PD-1 knockout mice.
  2. Although there are not data on the presence of pembrolizumab in either animal or human milk or its effects on breastfed children or on milk production, there is a potential for serious adverse reactions in breastfed children. Thus, women are advised not to breastfeed during treatment with pembrolizumab and for 120 days after the final dose.
* Patients with disease amenable to curative intent surgery.
* Patient has had a prior monoclonal antibody for treatment of sarcoma, unless the current regimen is checkpoint inhibitor immunotherapy.
* Patient has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin.
* Patient has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Patients with resolved childhood asthma, hypothyroidism stable on hormone replacement, Sjogren's syndrome, or with vitiligo would not be excluded. Patients requiring intermittent bronchodilators, inhaled steroids, or local steroid injections would not be excluded. Patients requiring physiologic doses of corticosteroids may be approved after consultation with the protocol principal investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility, measured as the number of patients completing treatment. | Up to 3 years
  Number of patients completing treatment with at least one cycle of pembrolizumab and completion of RT (Arm A) or completion of RT (Arm B). Up to 6 replacements are allowed (total subjects 6-12)

SECONDARY OUTCOMES:
Overall response rate (ORR) at non-irradiated sites | Up to 3 years.
  The overall response rate (ORR) at non-irradiated sites will be measured by iRECIST and will exclude the irradiated tumor. ORR rate is defined as the number of patients with a best overall response (BOR/iBOR) of complete response (CR/iCR) or partial response (PR/iPR) divided by the total number of patients enrolled in the study.
Local failure at the irradiated site | Up to 3 years
  Local failure rate at the irradiated site will be determined using cumulative incidence rates with death as a competing event at 12 months after initiation of treatment
Duration of response | Up to 3 years
  The duration of response is measured from the time measurement criteria are met for CR/PR or iCR/iPR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Progression-free survival | Up to 3 years.
  Progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Estimates at 6 and 12 months will be made.
Overall survival | Up to 3 years
  The duration of time from start of treatment to time of progression or death, whichever occurs first. Estimates at 6 and 12 months will be made.
Number of grade 3-5 adverse events | Up to 3 years.
  Severe toxicity will be measured by cumulative CTCAE v5.0 grade 3-5 events. Evaluation for toxicity will be made at Day 1 of each cycle, end of treatment, and in follow-up for up to 12 months following discontinuation of treatment.
Patient reported health-related quality of life | Up to 3 years.
  Mean summary score of the Functional Assessment of Cancer Therapy-General (FACT-G)
Patient reported toxicity | Up to 3 years.
  Mean summary score of the Functional Assessment of Cancer Therapy-Immune Checkpoint Modulator (FACT-ICM).
Patient reported treatment satisfaction | Up to 3 years.
  Mean summary score of the Functional Assessment of Chronic Illness Therapy-Treatment Satisfaction-General (FACIT-TS-G).

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Harris, MD, MPhil, Principal Investigator — University of California, Irvine
Locations (1):
- Chao Family Comprehensive Cancer Center, University of California, Irvine, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harris JP, Park J, Ku E, Seyedin S, Stitzlein R, Goldin A, Chen WP, McLaren C, Chen AM, Chow W. A Pilot Study of Pembrolizumab Combined With Stereotactic Ablative Radiotherapy for Patients With Advanced or Metastatic Sarcoma. Cancer Control. 2024 Jan-Dec;31:10732748241237331. doi: 10.1177/10732748241237331. PMID 38449377